CLINICAL TRIAL: NCT03838770
Title: Transcranial Direct Current Stimulation (tDCS) for the Management of Multiple Sclerosis Related Fatigue
Brief Title: tDCS for the Management of Multiple Sclerosis Related Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-01406
Record Dates: First submitted 2019-02-11; First posted 2019-02-12 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental)
  Interventions: Device: Active tDCS
- Sham (Placebo Comparator)
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: Active tDCS — Active target 2.0mA tDCS (n=60)
  Other Names: Soterix Mini-Ct Device
  Arms: Active
Device: sham tDCS — sham left-anodal dorsolateral prefrontal cortex (DLFPC) montage
  Arms: Sham

SUMMARY:
This is a pragmatic clinical trial that aims to determine the effect of tDCS on symptomatic fatigue in Multiple Sclerosis (MS) patients. This is a randomized, blinded, sham-controlled study design to determine the effect of Transcranial Direct Current Stimulation (tDCS) on MS participants to reduce feelings of fatigue.120 participants with MS and clinically-significant fatigue (as defined by a score of >36 on the Fatigue Severity Scale) will be recruited to participate in either an active or sham treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Definite MS diagnosis, all subtypes
* Fatigue Severity Scale score of 36 or greater
* Score of 7.5 or less on the Expanded Disability Status Scale (EDSS) (with caregiver proxy required for those with scores of 7.5 or greater)
* Ability to understand the informed consent process and provide consent to participate in the study

Exclusion Criteria:

* Primary neurologic, psychiatric or other medical disorder other than MS
* History of seizures or seizure disorder
* History of head trauma or medical device in head or neck
* Clinically significant abnormality on EKG
* Current symptomatic treatment for fatigue
* Symbol Digit Modalities Test or SDMT score≥3.0 SD from published norms
* WRAT-4 reading level below average (<85) (estimated general intellectual function)
* Beck Depression Inventory-Fast Screen (BDI- FS) score ≥10
* Current chronic headaches or migraines
* Skin disorder/sensitive near stimulation locations

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
change from baseline in the self-reported Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue instrument. | 7 Days post end of Treatment
  The minimally important difference representing a clinically significant improvement in patient-reported fatigue on the 7-item PROMIS Fatigue Scale is defined as a 3.0 point change in raw score. Clinically-significant response to tDCS treatment by the conservative measurement of >3.0 points on the PROMIS Fatigue Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: For individual participant data meta-analysis. Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.

REFERENCES:
- [Derived] Charvet L, Goldberg J, Li X, Best P, Shaw M, Ryerson LZ, Gutman J, Bikson M, Pilloni G, Krupp L. Enhanced cognitive outcomes with telehealth-based tDCS in multiple sclerosis: Results from a sham-controlled RCT. Mult Scler J Exp Transl Clin. 2025 Jul 28;11(3):20552173251356704. doi: 10.1177/20552173251356704. eCollection 2025 Jul-Sep. PMID 40735472